CLINICAL TRIAL: NCT06320782
Title: Effects of Different Dietary Interventions on Abdominal Fat Components, Quadriceps Muscles and Cardiometabolic Parameters: a Randomized Clinical Trial
Brief Title: Effects of Different Dietary Interventions on Abdominal Fat Components, Quadriceps Muscles and Cardiometabolic Parameters
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Isa Galvão Rodrigues, Principal Investigator, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4659262
Record Dates: First submitted 2024-01-17; First posted 2024-03-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Abdominal Obesity; Cardiac Disease; Metabolic Disease; Cardiometabolic Syndrome; Sarcopenia
Keywords: Cardiometabolic Risk Factors; Dietetic interventions; Abdominal Obesity; sarcopenia
MeSH Terms: conditions — Obesity, Abdominal; Heart Diseases; Metabolic Diseases; Metabolic Syndrome; Sarcopenia | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: 4 interventions distributed in a randomized manner among 4 different groups
Who Masked: Outcomes Assessor
Masking Description: The data analysis and interpretation stage will be carried out by the study coordinator, who will not have knowledge about the allocation of participants among the intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary intervention 1 (Experimental): Calorie restriction and balanced distribution of macronutrients
  Interventions: Behavioral: Calorie restriction and balanced distribution of macronutrients
- Dietary intervention 2 (Experimental): Calorie restriction and low-carbohydrate diet
  Interventions: Behavioral: Calorie restriction and low-carbohydrate diet
- Dietary intervention 3 (Experimental): Calorie restriction and low-fat diet
  Interventions: Behavioral: Calorie restriction and low-fat diet
- Dietary intervention 4 (Experimental): Collective nutritional guidance
  Interventions: Behavioral: Collective nutritional guidance

INTERVENTIONS:
Behavioral: Calorie restriction and balanced distribution of macronutrients — Progressive reduction of 500 to 1000 calories from the usual food intake or the recommendation of 20 calories/kg of current weight/day and distribution of macronutrients: 5% of carbohydrates, 2% of proteins and 3% of fats
  Arms: Dietary intervention 1
Behavioral: Calorie restriction and low-carbohydrate diet — Reduction in carbohydrate consumption and an increase in fat and protein intake, with the following proportions: 45% fat, 20% protein and 35% carbohydrate
  Arms: Dietary intervention 2
Behavioral: Calorie restriction and low-fat diet — Restriction of fat consumption and an increase in carbohydrate consumption, with the following proportions: 20% fat, 15% protein and 65% carbohydrate
  Arms: Dietary intervention 3
Behavioral: Collective nutritional guidance — Recommendations of the Food Guide for the Brazilian Population: limitation of the intake of foods with high energy density from fats and simple carbohydrates; substitution of saturated fats for unsaturated fats; exclusion of trans fat from the diet; increasing fruit and vegetable consumption to a daily minimum of 400g; increased consumption of high-fibre foods and limiting the consumption of sugars and salt.
  Arms: Dietary intervention 4

SUMMARY:
The study aims to evaluate the impact of different dietary interventions on body composition (abdominal fat components and quadriceps muscles) and cardiometabolic parameters. This is a randomized clinical trial study conducted in overweight adults, selected by voluntary adherence, in an outpatient clinic of a cardiology hospital. The sample was calculated based on data from a study with the Brazilian population, with the sample size calculated as a function of a mean difference (d) in visceral adipose tissue (VAT) after the interventions, standard deviation (s) and a significance level of 5% (z). To correct eventual losses, the number was increased by 20%. Four dietary interventions will be applied in the 6-month period: group with calorie restriction and balanced distribution of macronutrients (group 1); group with calorie restriction and low-carbohydrate diet (group 2); group with calorie restriction and low-fat diet (group 3) and group with collective nutritional guidance (group 4). Patients will be followed up monthly for the first 6 months to assess weight loss, analyze adherence to the diet therapy plan, reinforce nutritional guidelines, and monitor anthropometric measurements, abdominal adipose tissue, quadriceps muscles, and biochemical parameters. A reassessment will be performed at 12 months to analyze weight regain, analysis of anthropometric measurements, abdominal adipose tissue, quadriceps musculature and biochemical parameters. The evaluation of VAT, subcutaneous adipose tissue (SAT) and quadriceps musculature by ultrasound will be performed at baseline and after 3, 6 and 12 months of intervention. The present study is expected to clarify the effects that different dietary interventions produce over 3, 6 and 12 months on weight, abdominal fat deposits, quadriceps muscles and cardiometabolic parameters.

DETAILED DESCRIPTION:
The study aims to evaluate the impact of different dietary interventions on abdominal fat components, quadriceps musculature and cardiometabolic parameters. This is a randomized clinical trial study conducted in overweight adults, selected by voluntary adherence, in an outpatient clinic of a cardiology hospital. The sample will take place by voluntary adherence, after evaluation of the eligibility criteria and signing of the Free and Informed Consent Form. The sample was calculated based on data from a study with the Brazilian population , with the sample size calculated calculated as a function of a mean difference between the initial visceral adipose tissue (VAT) concentration and after dietary intervention, obtaining a minimum sample of 100 individuals. To correct eventual losses, this number was increased by 20%, totaling a sample n of 120 individuals. Four dietary interventions will be applied: group with calorie restriction and balanced distribution of macronutrients (group 1), considering a progressive reduction of 500 to 1000 calories from the usual food intake or the recommendation of 20 calories/kg of current weight/day and distribution of macronutrients: 5% of carbohydrates, 2% of proteins and 3% of fats; group with calorie restriction and low-carbohydrate diet (group 2), considering a reduction in carbohydrate consumption and an increase in fat and protein intake, with the following proportions: 45% fat, 20% protein and 35% carbohydrate ; group with calorie restriction and low-fat diet (group 3), considering a restriction of fat consumption and an increase in carbohydrate consumption, with the following proportions: 20% fat, 15% protein and 65% carbohydrate and group with collective nutritional guidance (group 4), considering the recommendations of the Food Guide for the Brazilian Population. Patients will be followed up monthly for the first 6 months to assess weight loss, analyze adherence to the diet therapy plan, reinforce nutritional guidelines, and monitor anthropometric measurements, abdominal adipose tissue, quadriceps muscles, and biochemical parameters. A reassessment will be performed at 12 months to analyze weight regain, analysis of anthropometric measurements, abdominal adipose tissue, quadriceps musculature and biochemical parameters. The evaluation of VAT, subcutaneous adipose tissue (SAT) and quadriceps musculature by ultrasound will be performed at baseline and after 3, 6 and 12 months of intervention. The weight loss will be evaluated as a percentage (%), based on the difference between the weight at the outcome and the weight at baseline. The weight regain will be calculated considering the difference between weight at outcome (at 6 months) and weight after six months of completion of the dietary intervention (at 12 months from the start of the study). The following parameters will be monitored: blood pressure, biochemical tests (leptin, adiponectin, fasting glucose, fasting insulin, glycated hemoglobin, triglycerides, total cholesterol and fractions, and C-reactive protein), anthropometric measurements (weight, height, waist circumference, and abdominal circumference), demographic variables (age, gender, schooling) and socioeconomic status. Data will be analyzed using the Statistical Package for Social Sciences - version 13.0 . In the description of the proportions, the binomial distribution will be approximated to the normal distribution by the 95% confidence interval. The proportions will be compared by the Chi-square test. Student's t-tests for paired or Wilcoxon samples will be used to compare VAT, SAT, quadriceps musculature, weight, BMI and biochemical parameters before and after the intervention of each group. To compare the changes in VAT, SAT, quadriceps musculature, anthropometric and biochemical parameters between the intervention groups, the one way or Kruskal Wallis ANOVA test will be used. Statistical significance will be established when a p<0.05 value. The present study is expected to clarify the effects that different dietary interventions produce over 3, 6 and 12 months on weight, abdominal fat deposits, quadriceps muscles and cardiometabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes, aged ≥20 years, Body Mass Index (BMI) ≥25kg/m², attended at the general Nutrition outpatient clinic of a public university hospital reference in cardiology.

Exclusion Criteria:

* Malnourished and eutrophic individuals;
* Individuals with liver disease and/or splenomegaly, ascites, or with recent abdominal surgery;
* Pregnant women and women who had children up to 6 months prior to the survey screening;
* Individuals with consumptive diseases whose weight loss may be a consequence;
* Individuals with hypothyroidism or hyperthyroidism, on pharmacological therapy for weight loss and/or on hormone therapy;
* Individuals with mental or psychological illnesses that may make it difficult to understand dietary guidelines;
* Individuals with physical limitations that made it impossible to carry out the anthropometric and abdominal adipose tissue evaluations.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Thickness, measured in centimeters, of visceral adipose tissue and quadriceps muscles | 3,6 and 12 months
  The effects that different dietary interventions produce on visceral adipose tissue thickness and quadriceps muscles( measured en centimeters) will be evaluated
Weight loss measured in kilograms | 6 months
  The effect of different dietary interventions produce on weight, measured in kilograms, will be evaluated
Thickness of quadriceps muscle | 3,6 and 12 months
  Thickness, measured in centimeters, of quadriceps muscle

SECONDARY OUTCOMES:
Serum levels of fasting glucose | 6 months
  The effects that different dietary interventions produce in serum levels of fasting glucose ( in mg/dl).), will be evaluated.
Serum levels of Insulin | 6 months
  The effects that different dietary interventions produce in serum levels of insulin in Microinternational Unit per Milliliter (μIU/mL)), will be evaluated.
Serum levels Triglycerides | 6 months
  The effects that different dietary interventions produce in serum levels of triglycerides (in mg/dl), ), will be evaluated.
Serum levels Lipid profile | 6 months
  The effects that different dietary interventions produce in serum levels of cholesterol (in mg/dl) , low-density lipoprotein cholesterol (LDL-C) ( in mg/dl), high-density lipoprotein cholesterol (HDL-C) ( in mg/dl), ), will be evaluated.
Serum levels C-reactive protein (hs-CRP) | 6 months
  The effects that different dietary interventions produce in serum levels of C-reactive protein (hs-CRP) (in mg/dl)), will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Isa Galvao Rodrigues, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Souza RJ, Bray GA, Carey VJ, Hall KD, LeBoff MS, Loria CM, Laranjo NM, Sacks FM, Smith SR. Effects of 4 weight-loss diets differing in fat, protein, and carbohydrate on fat mass, lean mass, visceral adipose tissue, and hepatic fat: results from the POUNDS LOST trial. Am J Clin Nutr. 2012 Mar;95(3):614-25. doi: 10.3945/ajcn.111.026328. Epub 2012 Jan 18. PMID 22258266